CLINICAL TRIAL: NCT04694495
Title: HPV Infection and Genital Microecology of Childbearing-age Female in China: A Cohort and Multicenter Study
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Peking University First Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Hainan General Hospital (Other); LanZhou University (Other); Lianyungang Hospital Affiliated Bengbu Medical College (Other); General Hospital of Ningxia Medical University (Other); Jinan Central Hospital (Other); Tibet Autonomous Region People's Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Anhui Provincial Hospital (Other Government); The First People's Hospital of Zunyi (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); First Affiliated Hospital, Sun Yat-Sen University (Other); Zhuhai Center for Maternal and Child Health Care (Other); First Affiliated Hospital of Guangxi Medical University (Other); Qinghai Red Cross Hospital (Other); Changzhi People's Hospital (Other); Shanghai East Hospital (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Huizhou Municipal Central Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Yuebei People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Fujian Maternity and Child Health Hospital (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Henan Provincial People's Hospital (Other); The Fifth Affiliated Hospital of Southern Medical University (Other); Shandong Provincial Hospital (Other Government); First Hospital of China Medical University (Other); Gansu Provincial Hospital (Other)
Responsible Party: Principal Investigator, Muxuan Chen, Diagnostic Technician, Zhujiang Hospital
Other Study IDs: CALM2004
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Papillomavirus Infections; Uterine Cervical Neoplasms; Sexual Transmitted Disease
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen will include cervical and vaginal swabs, cervical exfoliated cells from reproductive tract of the volunteers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- volunteers from health examination center: volunteers(n = 50/center) doing gynecologial examination recruited from health examination center, who shows no symptoms and signs in reproductive tract and are potentially regarded as the healthy controls
  Interventions: Diagnostic Test: 16S rRNA gene sequencing of cervical secretions
- volunteers from gynecology outpatient: volunteers(n = 150/center) recruited from gynecology outpatient, who show abnormal symptoms and signs in reproductive tract and are potentially regarded as the cases with conditions in reproductive tract
  Interventions: Diagnostic Test: 16S rRNA gene sequencing of cervical secretions

INTERVENTIONS:
Diagnostic Test: 16S rRNA gene sequencing of cervical secretions — 1. 16S rRNA gene sequencing of vaginal secretions: using NGS technology to assess the microbiota of the vaginal secretions
  2. Microecology assessment of vaginal secretions: morphology test, functional assessment and Nugent score assessment of the vaginal secretions are included.
  3. Genotyping of HPV and detection of sexually transmitted diseases pathogens based on the cervical exfoliated cells
  4. Thinprep cytologic test of cervical exfoliated cells: to evaluate the grade of cervical intraepithelial neoplasia
  Other Names: Microecology assessment of cervical secretions; Genotyping of HPV and detection of sexually transmitted diseases pathogens; Thinprep cytologic test of cervical exfoliated cells

SUMMARY:
The purpose of this study to access the relations between genital microecology, HPV infection and cervical intraepithelial neoplasia of childbearing-age female in China

DETAILED DESCRIPTION:
The volunteers will be recruited from the women who come to the hospital to do the thinprep cytologic test. After being informed about the potential risks, each volunteer giving written informed consent will be asked to complete a questionnaire. Then, cervical and vaginal swabs and cervical exfoliated cells will be taken from each volunteer to perform 16S rRNA gene sequencing microecology assessment on cervical secretions and detection and genotyping of HPV and pathogens of sexually transmitted diseases. If there is something abnormal with the diagnostic outcomes in the previous examinations, according to the doctor's judgement, those volunteer will be asked to undergo a vaginoscope and a cervical biopsy to evaluate the grade of cervical intraepithelial neoplasia. After six months since the entry, each volunteer will be asked to go back to each research center to do the same sampling and examination as previously did in entry.

ELIGIBILITY:
Inclusion Criteria:

* Female of childbearing age conducting thinprep cytologic test
* Having an experience of sexual intercourse
* Not during the menstrual period
* No sexual intercourse or vaginal medication or vaginal flushing in 3 days before sampling

Exclusion Criteria:

* Within 8 weeks of pregnancy or postpartum
* Having had tumors in reproductive tract
* Having had HPV bivalent, tetravalent or nine-valent vaccination
* Having received treatment for anti- HPV or other STDs pathogens infection
* Having had hysterectomy, cervical surgery and pelvic radiotherapy
* Having used broad-spectrum antibiotics, probiotics or vaginal suppositories in reproductive tract within 1 month

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers will be recruited from both outpatient department of gynecology and health examination center in each research center
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
alteration of genital microecology from baseline at month 6 | basline and month 6
  Genital microecology includes measurements of cervical microbiota, HPV and other sexually transmitted diseases pathogens infection status, conditions of the vaginal secretion and the grade of cervical intraepithelial neoplasia. As for cervical microbiota, the NGS technology will be used to sequence the 16s rRNA gene of the microbes in the cervical secretion of each volunteers. PCR will be used to detect HPV and other sexually transmitted diseases pathogens. As for the conditions of the vaginal secretion, methods such as manual microscopic inspection, gram stain and enzymology test will be used to do the measurement. Moreover, thinprep cytologic test of cervical exfoliated cells will be performed to evaluate the grade of cervical intraepithelial neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Doctor, Principal Investigator — Department of Laboratory Medicine, Zhujiang Hospital, Southern Medical University
Locations (42):
- China (42):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Chaozhou Central Hospital, Chaozhou, Guangdong
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong Provincial Hospital of Intergrated Traditional Chinese and Western Medicine, Foshan, Guangdong
  - Zhujiang Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Taihe Branch of Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Hospital of Guangzhou University of Chinese Medicine, Shenzhen, Guangdong
  - Shenzhen Luohu Hospital Group Luohu People's Hospital, Shenzhen, Guangdong
  - The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Xiaolan People's Hospital of Zhongshan, Zhongshan, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen Univeristy, Guangzhou, Guangzhou
  - Zhuhai Women and Children's Hospital, Zhuhai, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First People's Hospital of Zunyi, Zunyi, Guizhou
  - Yue Bei People's Hospital, Shaoguan, Gunagdong
  - Hainan General Hospital, Haikou, Hainan
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital fo Qiqihar, Qiqihar, Hei Longjiang
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Jilin Central General Hospital, Jilin, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai Red Cross Hospital, Xining, Qinghai
  - Jinan Central Hospital, Jinan, Shandong
  - Obstetrics&Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tibet Autonomous Region People's Hospital, Lhasa, Tibet
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hanzhou, Zhejiang
  - Changsha Central Hospital, Changsha
  - The Third Affiliated Hospital of CQMU, Chongqing
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Shanghai East Hospital Tongji University, Shanghai

REFERENCES:
- [Derived] Chen M, Qi C, Qing W, Zhou Z, Zhang Y, Chen R, Hou Y, Ou J; CALM2004 Consortium Investigators; He Y, Zhou H. Vaginal microbiome and sexually-transmitted pathogens in Chinese reproductive-age women: a multicentre cross-sectional and longitudinal cohort study. Nat Commun. 2025 Nov 14;16(1):10002. doi: 10.1038/s41467-025-64917-7. PMID 41238551
- [Derived] Zhang Y, Qing W, Mo W, Chen R, Zhou Z, Hou Y, Shi Y, Qi C, Ou J, Xie L; CALM 2004 Study Group; Wang Y, Zhou H, Chen M. U. Parvum serovars exhibit distinct pathogenicity in Chinese women of childbearing age: a multicentre cross-sectional study. BMC Infect Dis. 2024 Oct 28;24(1):1213. doi: 10.1186/s12879-024-10113-9. PMID 39468466